CLINICAL TRIAL: NCT04668144
Title: Pharmacodynamic and Pharmacokinetic Profiles on Switching From Cangrelor to Prasugrel in Patients With Acute Coronary Syndrome Undergoing Percutaneous Coronary Intervention: The Switching Antiplatelet -6 (SWAP-6) Study
Brief Title: Pharmacodynamic and Pharmacokinetic of Switching From Cangrelor to Prasugrel in ACS Patients Undergoing PCI
Acronym: SWAP-6
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Scott R. MacKenzie Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMF-02
Record Dates: First submitted 2020-12-09; First posted 2020-12-16 (Actual); Results first posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Coronary Artery Disease; Acute Coronary Syndrome
MeSH Terms: conditions — Coronary Artery Disease; Acute Coronary Syndrome | interventions — cangrelor; Prasugrel Hydrochloride

STUDY DESIGN:
Masking Description: Laboratory personnel will be blinded to treatment assignments
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Prasugrel (Active Comparator): Prasugrel only administered at the start of PCI
  Interventions: Drug: Prasugrel
- Prasugrel + Cangrelor (Experimental): Cangrelor plus prasugrel concomitantly administered at the start of PCI
  Interventions: Drug: Cangrelor; Drug: Prasugrel
- Cangrelor followed by Prasugrel (Active Comparator): Cangrelor administered at the start of PCI plus prasugrel administered at the end of the cangrelor infusion
  Interventions: Drug: Cangrelor; Drug: Prasugrel

INTERVENTIONS:
Drug: Cangrelor — Cangrelor will be used at the FDA recommended dose using a 30 μg/kg bolus followed by 4 μg/kg/min infusion. The total infusion will last 2 hours.
  Other Names: Kengreal
  Arms: Cangrelor followed by Prasugrel; Prasugrel + Cangrelor
Drug: Prasugrel — Prasugrel will be used in line with FDA recommendations using a 60mg LD followed by a 10mg daily maintenance dose started 24 hours after LD administration
  Other Names: Effient

SUMMARY:
Cangrelor is an intravenous P2Y12 inhibitor utilized as a bridge to achieve adequate platelet inhibition until oral P2Y12 inhibitors achieve their full antiplatelet effects in patients undergoing coronary stenting. Although in this setting the potent oral P2Y12 inhibitor prasugrel is commonly utilized, there is very limited data on the optimal approach for switching between these therapies. The overarching aim of this investigation is to rule out a drug drug interaction (DDI) when cangrelor and prasugrel are concomitantly administered in patients undergoing coronary stenting.

DETAILED DESCRIPTION:
Cangrelor is an intravenous P2Y12 inhibitor utilized as a bridge to achieve adequate platelet inhibition until oral P2Y12 inhibitors achieve their full antiplatelet effects in patients undergoing coronary stenting. Although in this setting the potent oral P2Y12 inhibitor prasugrel is commonly utilized, there is very limited data on the optimal approach for switching between these therapies. In particular, ruling out a drug-drug interaction (DDI) is critical to this extent as the presence of a DDI would translate into reduced or abolished antiplatelet effects exposing these acute patients to an increased thrombotic risk. There is an unmet need to better elucidate pharmacodynamic profiles associated with the transition from cangrelor to prasugrel therapy. Of note, prasugrel has recently gone off patent and the availability of a generic formulation will favorably impact its use. Pharmacodynamic studies provide some support on the safety of administering prasugrel at the start of cangrelor infusion. However, the available data does not allow to rule out a DDI given that there was no comparator arm in which prasugrel was either given alone or at the end of cangrelor infusion. The methodological approach for this assessment should rely on comprehensive pharmacodynamics investigations aimed to assess levels of P2Y12 receptor inhibition, pharmacokinetic investigations to assess systemic levels of the drug/drug metabolite, and mechanistic investigations by assessment of levels of P2Y12 receptor gene expression. The overarching aim of this investigation is to rule out a DDI when cangrelor and prasugrel are concomitantly administered in patients undergoing coronary stenting.

ELIGIBILITY:
Inclusion Criteria:

* Patients with NSTE-ACS (UA or NSTEMI) undergoing PCI. NSTE-ACS will be defined as the presence of cardiac ischemic symptoms with ischemic changes (but not ST-segment elevation) on electrocardiogram with or without a positive troponin. However, normal electrocardiograms will be acceptable if the investigator will consider an ACS presentation likely.
* Age between 18 and 75 years old

Exclusion Criteria:

* Inability to provide written informed consent
* Age >75 years
* Weight <60 Kg
* ST-segment elevation myocardial infarction
* On treatment with a P2Y12 receptor antagonist (ticlopidine, clopidogrel, prasugrel, ticagrelor) in past 7 days
* Known allergies to prasugrel or cangrelor
* Considered at high risk for bleeding
* History of ischemic or hemorrhagic stroke or transient ischemic attack
* On treatment with oral anticoagulant (Vitamin K antagonists, dabigatran, rivaroxaban, apixaban, edoxoban)
* Planned treatment with glycoprotein IIb/IIIa inhibitors (only bailout use allowed)
* Fibrinolytics within 24 hours
* Known platelet count <80x106/mL
* Known hemoglobin <10 g/dL
* Active bleeding
* Known end stage renal disease on hemodialysis
* Known severe hepatic dysfunction
* Intubated patients (prior to randomization)
* Pregnant females [women of childbearing age must use reliable birth control (i.e. oral contraceptives) while participating in the study]

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 359 (Actual)
Dates: Start 2021-02-18 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2023-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Franchi, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida Jacksonville, Jacksonville, Florida, United States

REFERENCES:
- [Derived] Franchi F, Rollini F, Ortega-Paz L, Been L, Giordano S, Galli M, Ghanem G, Garabedian H, Al Saleh T, Uzunoglu E, Rivas A, Pineda AM, Suryadevara S, Soffer D, Zenni MM, Mahowald M, Reiter B, Jilma B, Angiolillo DJ. Switching From Cangrelor to Prasugrel in Patients Undergoing Percutaneous Coronary Intervention: The Switching Antiplatelet-6 (SWAP-6) Study. JACC Cardiovasc Interv. 2023 Oct 23;16(20):2528-2539. doi: 10.1016/j.jcin.2023.08.009. Epub 2023 Aug 21. PMID 37609698

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between February 18, 2021 and February 2, 2023, 359 patients provided written informed consent to participate in the study
Pre-assignment Details: 282 patients were excluded because they had at least one exclusion criteria.
Period: Overall Study
Arm/Group | Prasugrel | Prasugrel + Cangrelor | Cangrelor Followed by Prasugrel
Started | 25 | 25 | 27
Completed | 25 | 24 | 25
Not Completed | 0 | 1 | 2
Not completed — Protocol Violation | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Population: Patients who were randomized and received study medications
Groups:
- Total: Total of all reporting groups
Arm/Group | Prasugrel | Prasugrel + Cangrelor | Cangrelor Followed by Prasugrel | Total
Number analyzed (Participants) | 25 | 25 | 27 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (9) | 64 (8) | 63 (8) | 63 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 7 | 7 | 17
  Male | 22 | 18 | 20 | 60
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 1 | 7 | 13
  White | 20 | 21 | 18 | 59
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 2 | 3
Acute coronary syndrome [Count of Participants; unit: Participants] | 9 | 10 | 10 | 29

OUTCOME MEASURES:

1. Primary Outcome: Platelet Reactivity Measured by VerifyNow
Description: The primary end point of the study will be the non-inferiority in P2Y12 reaction units (PRU) of cangrelor plus prasugrel concomitantly administered at the start of PCI versus prasugrel only administered at the start of PCI.
Time Frame: 4 hours
Population: Patient with valid primary end point data
Measure: Mean (Standard Deviation); unit: PRU
Arm/Group | Prasugrel | Prasugrel + Cangrelor | Cangrelor Followed by Prasugrel
Number analyzed (Participants) | 24 | 24 | 24
PRU | 23 (31) | 153 (104) | 65 (84)
Statistical Analysis 1: Comparison: Prasugrel vs Prasugrel + Cangrelor; The primary hypothesis of our study was that in patients receiving concomitant administration of cangrelor and prasugrel (experimental arm), platelet inhibition as assessed by PRU would be noninferior to patients receiving prasugrel only (active control); Test type: Non-Inferiority — Under the assumption of 0 difference in mean PRU between groups and a common standard deviation of 50 PRU, a sample size of 22 patients per group would allow for the 95%CI to stay within ± 45 PRU with a 90% power and alpha=0.05. In line with previously reported investigations, 45 PRU was chosen for the noninferiority margin for the upper 95%CI limit of the difference; ANCOVA — p-value was not calculated for noninferiority analysis; Mean Difference (Final Values) = 130, 95% CI 2-sided [85 to 176]

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | Prasugrel | Prasugrel + Cangrelor | Cangrelor Followed by Prasugrel
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 2/27
Other Adverse Events (participants affected / at risk) | 8/25 | 2/25 | 4/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prasugrel (N=25) | Prasugrel + Cangrelor (N=25) | Cangrelor Followed by Prasugrel (N=27)
Asystole (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — Asystole after nitroglycerine given in Cath lab
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) — Acute respiratory failure requiring intubation during procedure
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prasugrel (N=25) | Prasugrel + Cangrelor (N=25) | Cangrelor Followed by Prasugrel (N=27)
Minor bleeding (Blood and lymphatic system disorders) | 8 (8) | 2 (2) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-05-03): https://cdn.clinicaltrials.gov/large-docs/44/NCT04668144/Prot_SAP_000.pdf
  • Informed Consent Form (2020-12-11): https://cdn.clinicaltrials.gov/large-docs/44/NCT04668144/ICF_001.pdf